CLINICAL TRIAL: NCT01378221
Title: Vitamin D Metabolism in Senescent Cardiac Surgery Patients
Acronym: VISE
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: 005
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Bypass Grafting; Heart Valve Surgery
Keywords: vitamin D; cardiac surgery; inflammation; immune system; age
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: cardiac surgery patients age 65 years and less
- Group 2: cardiac surgery patients aged 75 years and over

SUMMARY:
Advanced age is associated with an increase in postoperative morbidity and mortality in cardiac surgery patients. In detail, compared with younger patients those aged 75 years and older have significantly higher rates of in-hospital mortality, cerebrovascular events, pneumonia, and dialysis. In addition, older cardiac surgery patients have longer mechanical ventilation times. Vitamin D exerts several beneficial effects on the cardiovascular system. Moreover, it has immuno-modulatory and anti-inflammatory properties. The hormonal form of vitamin D, 1,25-dihydroxyvitamin D, is an independent predictor of mid-term mortality in cardiac transplant recipients. 1,25-dihydroxyvitamin D also predicts mid-term and long-term mortality in patients with a high risk for cardiovascular disease. Mild renal impairment, insufficient vitamin D levels, and secondary hyperparathyroidism are common in frail elderly individuals. The present study aimed to investigate whether cardiac surgery exerts age-dependent effects on calciotropic hormones, components of the immune system, and inflammatory processes.It is hypothesized that (i) baseline 1,25-dihydroxyvitamin D levels are lower in patients <= 75 years of age compared to younger patients, (ii) cardiac surgery results in a transient decrease in circulating 1,25-dihydroxyvitamin D, and (iii) that the decrease in 1,25-dihydroxyvitamin D is probably more pronounced in older than in younger cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* age: <= 65 years and >= 75 years
* first elective cardiac surgery (bypass or combined bypass and heart valve surgery)
* written informed consent

Exclusion Criteria:

* emergency cardiac intervention
* primary hyperparathyreoidism
* primary and secondary hypoparathyreoidism
* daily vitamin D supplementation > 10 micrograms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elective cardiac surgery patients receiving isolated coronary artery bypass grafting or combined coronary artery bypass grafting and heart valve surgery
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Börgermann, MD, Principal Investigator — Heart Center NRW, Ruhr University Bochum, 32545 Bad Oeynhausen, Germany
Locations (1):
- Heart Center North Rhine-Westphalia, Bad Oeynhausen, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Borgermann J, Lazouski K, Kuhn J, Dreier J, Schmidt M, Gilis-Januszewski T, Knabbe C, Gummert JF, Zittermann A. 1,25-Dihydroxyvitamin D fluctuations in cardiac surgery are related to age and clinical outcome*. Crit Care Med. 2012 Jul;40(7):2073-81. doi: 10.1097/CCM.0b013e31824e8c42. PMID 22584760

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 36 | 39
Completed | 29 | 30
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 58.8 (5.92) | 77.0 (4.38) | 68.05 (5.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 27 | 21 | 48
Region of Enrollment [Number; unit: participants]
  Germany | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Peri- and Postoperative Time Course of Circulating 1,25-dihydroxyvitamin D in the First Postoperative Month in Cardiac Surgery Patients
Time Frame: change from baseline within 1 month after cardiac surgery
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 29 | 30
percentage | 13 (1.1) | 4.2 (0.2)

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No